CLINICAL TRIAL: NCT04121728
Title: Evaluation of the Modulation of Attention Explored in ERPs as a Marker of Early Cognitive Decline: Concept Validation on the Effect of Ginkgo Biloba Extracts. Randomized, Double-blind, Cross-over, Placebo-controlled Study
Brief Title: Modulation of Attention in Event Related Potential (ERPs) as a Marker of Early Cognitive Decline by Ginkgo Biloba
Acronym: AgilGinkgo
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jean-François Démonet (Other)
Collaborators: University of Lausanne Hospitals (Other)
Responsible Party: Sponsor-Investigator, Jean-François Démonet, Professor, MD.PhD, University of Lausanne Hospitals
Organization: University of Lausanne Hospitals (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2018-02134 BASEC
Record Dates: First submitted 2019-09-18; First posted 2019-10-10 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Subjective Cognitive Decline; Cognitive Performance; Functional Capacity; Age-related Cognitive Decline
Keywords: metrological characteristics of EEG-ERP; Ginkgo Biloba
MeSH Terms: interventions — Ginkgo biloba extract

STUDY DESIGN:
Intervention Model Description: randomized double-blind crossover design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigational Medicinal Product (IMP), e.g Placebo and Ginkgo Biloba, is located and dispensed by Central Pharmacy.
  Only pharmacists are not blinded but they are neither involved in the conduct of the study not the analysis of the results
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Ginkgo-Placebo (Other): Cross-over design: In Group Ginkgo-Placebo participants are allocated first to the IMP Symfona® during 6 months and after 2 months of wash-out period are allocated to the placebo for 6 months.
  Interventions: Drug: Ginkgo biloba extract; Drug: Placebo
- Group Placebo-Ginkgo (Other): Cross-over design:In Group Placebo-Ginkgo participants are allocated first to the placebo during 6 months and after 2 months of wash-out period are allocated the IMP Symfona® for 6 months.
  Interventions: Drug: Ginkgo biloba extract; Drug: Placebo

INTERVENTIONS:
Drug: Ginkgo biloba extract — Symfona® commercial standardized Ginkgo biloba extracts are used in this study, at a rate of 2 capsules of 120 mg per day for 170 days.
  Other Names: Symfona®
Drug: Placebo — The placebo is presented in the form of capsules of identical mass, color and shape to those of the study product. It is composed of lactose, the excipients present in Symfona® 120 mg and colorants. The dosage is identical to that of the investigational product.
  Other Names: Placebo caps

SUMMARY:
The objective of this study is to simultaneously establish the metrological characteristics of the new executive function markers (decision making and multiple flow management) derived from repeated ERP variations and to identify their ability to test whether a short treatment using Ginkgo biloba versus placebo extracts can modify the cognitive performance and functional capacity of patients in the very early stages of age-related cognitive decline. This trial, using subjects as their own control (cross-over) in repeated measurements will establish the reproducibility characteristics of the measurements and intra-individual variations of ERP over time in this population

DETAILED DESCRIPTION:
This study is a single-center, randomized clinical trial testing the effects of Ginkgo biloba extracts versus placebo on event related potential ERP registration measurements in Electroencephalography (EEG) during neuropsychological tasks. The Hold-Release (HR) neuropsychological test allows the study of behavioral and neurofunctional correlates using several different techniques for online recording of brain activity. This test measures the engagement of focused attention and the loading of information into working memory, as opposed to the disengagement of attention.

The study will be carried out in a randomized cross-over design, with "Ginkgo" vs. Placebo", or inversely, for 170 days each (approximately 6 months), separated by an 8-weeks wash-out period. A follow-up visit will be held 3 months after the last treatment of the study.

The cross-over design uses each patient as its own control, which allows an easy comparison between the 2 groups "Placebo" vs. "Ginkgo" by limiting inter-patient variations. In addition, by doubling the number of patients per treatment compared to a classic study design in 2 groups, cross-over reduces the number of patients to be recruited, which facilitates recruitment on a single site.

The study requires the recruitment of sixteen (16) informative participants with cognitive complaints.

ELIGIBILITY:
Inclusion Criteria

* Signed consent form
* men and women
* 60 to 80 years old
* Diagnostic of Subjective complain
* Understanding the 2 Hold-Release tasks in ERP

Exclusion Criteria:

* Montreal Cognitive Evaluation Score (MoCA) <24
* Overall Clinical Dementia Rating (CDR) score > 0.5
* Scores of the Hospital Anxiety and Depression Scale (HADS): HADS-A (Anxiety) > 8 and/or HADS-D (Depression) > 8
* Mild Cognitive Impairment (MCI) or dementia
* Contraindication to MRI
* Atrophy of any region of the brain as seen in the T1 volumetric MRI sequence
* Any uncontrolled somatic or psychiatric condition
* Bleeding disorders, and/or taking medications that increase the risk of bleeding,
* Hypersensitivity to Ginkgo biloba or any of its excipients
* Lactose intolerance
* Treatment with barbiturates and/or neuroleptics
* Ongoing treatment with Ginkgo biloba derivatives (a period of 2 months without treatment before inclusion is required

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Reproducibility of contingent negative variation (CNV) event-related potential (ERP) component amplitude (microV) during the Hold-Release (HR) neuropsychological test | through study completion, an average of 14 months
  Reproducibility of CNV will be assessed by interclass correlation coefficient (ICC)
Intra-individual variability of contingent negative variation (CNV) event-related potential (ERP) component amplitude (microV) during the Hold-Release (HR) neuropsychological test | through study completion, an average of 14 months
  Intra-individual variability of CNV will be assessed by Interclass Coefficient Correlation (ICC)
Reproducibility of P300/P300' event-related potential (ERP) component amplitude (microV) during the Hold-Release (HR) neuropsychological test | through study completion, an average of 14 months
  Reproducibility of P300/P300' will be assessed by Interclass Coefficient Correlation (ICC)
Intra-individual variability of P300/P300' event-related potential (ERP) component amplitude (microV) during the Hold-Release (HR) neuropsychological test | through study completion, an average of 14 months
  Intra-individual variability of P300/P300' will be assessed by Interclass Coefficient Correlation (ICC)
Change in cognitive performance as assessed by variation in amplitude (mivroV) of the CNV component measured during the Hold-Release (HR) neuropsychological test after 6 months of Ginkgo biloba treatment | through study completion, an average of 14 months
  the statistical model of repeated measurements of variance analysis will be used
Change in cognitive performance as assessed by variation in amplitude (mivroV) of the P300/P300' component measured during the Hold-Release (HR) neuropsychological test after 6 months of Ginkgo biloba treatment | through study completion, an average of 14 months
  the statistical model of repeated measurements of variance analysis will be used

SECONDARY OUTCOMES:
Change in cognitive performance as assessed using the Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) test after 6 months of Ginkgo biloba treatment | 6 months
  the statistical model of repeated measurements of variance analysis will be used
Change in scores of categorical semantic verbal fluency after 6 months of Ginkgo biloba treatment | 6 months
  the statistical model of repeated measurements of variance analysis will be used
Change in scores of verbal fluency letter instruction after 6 months of Ginkgo biloba treatment | 6 months
  the statistical model of repeated measurements of variance analysis will be used
Change in anxiety and depression as assessed using the Hospital Anxiety and Depression Scale (HAD-A/D) after 6 months of Ginkgo biloba treatment | 6 months
  the statistical model of repeated measurements of variance analysis will be used
Change in reaction time (ms) during the Hold-Release (HR) neuropsychological test after 6 months of Ginkgo biloba treatment | 6 months
  the statistical model of repeated measurements of variance analysis will be used
Magnitude of repetition effects (Test-retest Reliability, TTR) on the contingent negative variation (CNV) event-related potential (ERP) component during the Hold-Release (HR) neuropsychological test. | through study completion, an average of 14 months
  Combination of an analysis of variance (ANOVA) in repeated measurements and an analysis of variance (ANOVA) in correlation analysis will be used to assess respectively differences (microV) between measurement sessions and the existence of shared associations (correlation coefficient).
Magnitude of repetition effects (Test-retest Reliability, TTR) on P300/P300' event-related potential (ERP) component during the Hold-Release (HR) neuropsychological test. | through study completion, an average of 14 months
  Combination of an analysis of variance (ANOVA) in repeated measurements and an analysis of variance (ANOVA) in correlation analysis will be used to assess respectively differences (microV) between measurement sessions and the existence of shared associations (correlation coefficient).
Association (correlation coefficient) between a transversal measurement of VPN event-related potential (ERP) component during the Hold-Release (HR) neuropsychological test and the conventional verbal fluency scores. | through study completion, an average of 14 months
  a mixed linear model approach will be applied to assess prediction
Association (correlation coefficient) between a transversal measurement of P300/P300' event-related potential (ERP) component during the Hold-Release (HR) neuropsychological test and the conventional verbal fluency scores. | through study completion, an average of 14 months
  a mixed linear model approach will be applied to assess prediction
Association (correlation coefficient) between a transversal measurement of VPN event-related potential (ERP) component during the Hold-Release (HR) neuropsychological test and evolution of its own value during the participant's follow-up | through study completion, an average of 14 months
  a mixed linear model approach will be applied to assess prediction
Association (correlation coefficient) between a transversal measurement of P300/P300' event-related potential (ERP) component during the Hold-Release (HR) neuropsychological test and evolution of its own value during the participant's follow-up | through study completion, an average of 14 months
  a mixed linear model approach will be applied to assess prediction

OTHER OUTCOMES:
Predictive metrological characteristics of ERP modulation in term of its ability to detect a more sensitive cognitive variation than usual method | through study completion, an average of 14 months
  a mixed linear model approach will be applied to assess prediction
Predictive metrological characteristics of ERP modulation in term of its ability to detect a slope break during cognitive decline | through study completion, an average of 14 months
  a mixed linear model approach will be applied to assess prediction

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François Démonet, Prof, Principal Investigator — Universitary Lausanne Hospital
Locations (1):
- Centre Leenaards de la mémoire (CLM) CHUV, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amieva H, Le Goff M, Millet X, Orgogozo JM, Peres K, Barberger-Gateau P, Jacqmin-Gadda H, Dartigues JF. Prodromal Alzheimer's disease: successive emergence of the clinical symptoms. Ann Neurol. 2008 Nov;64(5):492-8. doi: 10.1002/ana.21509. PMID 19067364
- [Background] Luck T, Luppa M, Matschinger H, Jessen F, Angermeyer MC, Riedel-Heller SG. Incident subjective memory complaints and the risk of subsequent dementia. Acta Psychiatr Scand. 2015 Apr;131(4):290-6. doi: 10.1111/acps.12328. Epub 2014 Sep 9. PMID 25201166
- [Background] Thierry G, Doyon B, Demonet JF. ERP mapping in phonological and lexical semantic monitoring tasks: A study complementing previous PET results. Neuroimage. 1998 Nov;8(4):391-408. doi: 10.1006/nimg.1998.0371. PMID 9811557
- [Background] Martin CD, Thierry G, Demonet JF. ERP characterization of sustained attention effects in visual lexical categorization. PLoS One. 2010 Mar 25;5(3):e9892. doi: 10.1371/journal.pone.0009892. PMID 20361039
- [Background] Tan MS, Yu JT, Tan CC, Wang HF, Meng XF, Wang C, Jiang T, Zhu XC, Tan L. Efficacy and adverse effects of ginkgo biloba for cognitive impairment and dementia: a systematic review and meta-analysis. J Alzheimers Dis. 2015;43(2):589-603. doi: 10.3233/JAD-140837. PMID 25114079
- [Background] Kennedy DO, Scholey AB, Drewery L, Marsh VR, Moore B, Ashton H. Electroencephalograph effects of single doses of Ginkgo biloba and Panax ginseng in healthy young volunteers. Pharmacol Biochem Behav. 2003 Jun;75(3):701-9. doi: 10.1016/s0091-3057(03)00120-5. PMID 12895688